CLINICAL TRIAL: NCT07040579
Title: Transcatheter Bioabsorbable Occluder Closure for Outlet Ventricular Septal Defect: Safety, Effectiveness and Impact on Aortic Valve Function
Brief Title: Bioabsorbable Occluder for Outlet VSD: Safety and Aortic Valve Effects
Acronym: ABSORB-VSD
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: GXMU-VSDO-001
Record Dates: First submitted 2025-05-28; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Congenital Heart Defects; VSD
Keywords: transcatheter; bioabsorbable occluder; outlet VSD
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BioOccl-VSD: Patients with outlet ventricular septal defects undergoing transcatheter closure with bioabsorbable occluders.
  Interventions: Device: transcatheter closure of outlet VSDs with bioabsorbable occluders

INTERVENTIONS:
Device: transcatheter closure of outlet VSDs with bioabsorbable occluders — Transcatheter closure of outlet ventricular septal defects using a bioabsorbable occluder (Shape Memory Alloy Ltd, Shanghai, China). Implantation is performed via femoral/transthoracic approach under echocardiographic guidance following standard interventional protocols.

SUMMARY:
This study aims to evaluate the efficacy and safety of transcatheter bioabsorbable occluder closure in patients with outlet-type ventricular septal defect (outlet VSD), with a focus on assessing its impact on aortic valve function.

DETAILED DESCRIPTION:
Outflow-type ventricular septal defects (outlet VSDs) represent a challenging subset of congenital heart defects due to their association with progressive aortic valve prolapse and regurgitation. While surgical repair remains the gold standard, no reliable occluder has been available for transcatheter closure of this defect subtype.

The anatomical proximity of outlet VSDs to the aortic valve has historically limited transcatheter interventions. Conventional eccentric metal occluders require strict patient selection, typically being feasible only in cases with small defects and minimal aortic valve prolapse. Moreover, long-term concerns persist regarding metal devices' impact on aortic valve function.

Bioabsorbable occluders have been clinically available for perimembranous VSD closure. Their soft material properties minimize mechanical trauma to the aortic valve, while gradual resorption over time may eliminate permanent device-related complications. However, robust data regarding their efficacy, safety, and long-term impact on aortic valve function in outlet VSDs remain lacking.

This study aims to evaluate the short- and long-term outcomes of bioabsorbable occluder closure in outlet VSD patients, with a focus on defect closure rates and aortic valve function preservation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥1 year and weight ≥10 kg
* Outlet VSD without ventricular malalignment
* Maximal defect diameter ≤12mm with subaortic rim ≤1mm and no ≥mild aortic regurgitation by by transthoracic or transesophageal echocardiography
* Written informed consent

Exclusion Criteria:

* Outlet VSD with a fibrous postero-inferior rim
* Concurrent cardiac conditions requiring surgical correction
* Severe pulmonary hypertension (PVR > 5 WU, assessed by right heart catheterization )
* Intracardiac thrombus
* Pregnancy
* Active systemic infection within 1 month

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients diagnosed with outlet ventricular septal defects who undergo transcatheter closure with bioabsorbable occluders
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2032-09-30 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with procedural success | 12 months
  1. Occluder in correct anatomical position
  2. Absence of major adverse events (all-cause mortality, all stroke, myocardial infarction, or re-hospitalization for device/procedure-related causes) 3) Residual shunt ≤ 2 mm and aortic regurgitation ≤ trace evaluated by transthoracic or transesophageal echocardiography

SECONDARY OUTCOMES:
Number of participants with technical success | Intraprocedural
  Absence of mortality, correct positioning of the occluder into the proper anatomical location， aortic regurgitation≤ trace by transthoracic or transesophageal echocardiography
Number of participants with major adverse events | 12/24/60 months
  All-cause mortality, all stroke, myocardial infarction, re-hospitalization for device or procedure-related causes
Closure Efficacy | Intraprocedural, 72 hours post procedure, 1/3/6/12/24/60 months
  1）Successful closure: Rate of successful VSD closure (residual shunt ≤2 mm) assessed by transthoracic or transesophageal echocardiography.
  2) Complete closure: Rate of complete closure (no residual shunt) assessed by transthoracic or transesophageal echocardiography.
Aortic regurgitation severity | Baseline, Intraprocedural, 72 hours post procedure, 1/3/6/12/24/60 months
  Aortic regurgitation severity measured by transthoracic and/or transesophageal echocardiography. Assessment of aortic regurgitation severity according to current recommendations for valvular heart disease.
Pulmonary regurgitation severity | Baseline, Intraprocedural, 72 hours post procedure, 1/3/6/12/24/60 months
  Pulmonary regurgitation severity measured by transthoracic and/or transesophageal echocardiography. Assessment of pulmonary regurgitation severity according to current recommendations for valvular heart disease.
Left ventricular outflow tract (LVOT) velocity and pressure gradient | Baseline, Intraprocedural, 72 hours post procedure, 1/3/6/12/24/60 months
  Peak LVOT velocity (m/s) and maximum instantaneous pressure gradient (mmHg) measured by continuous-wave Doppler (CWD) echocardiography, using the simplified Bernoulli equation (ΔP = 4v²).
Right ventricular outflow tract （RVOT）velocity and pressure gradient | Baseline, Intraprocedural, 72 hours post procedure, 1/3/6/12/24/60 months
  Peak LVOT velocity (m/s) and maximum instantaneous pressure gradient (mmHg) measured by continuous-wave Doppler (CWD) echocardiography, using the simplified Bernoulli equation (ΔP = 4v²).
Disc area quantification | 72 hours post procedure, 1/3/6/12/24/60 months
  Left and right disc areas are measured by transthoracic echocardiography (TTE) planimetry in parasternal short-axis (PSAX), apical long-axis (ALAX), and apical 5-chamber (A5C) views using QLAB 3DQ Advanced software (Philips). The mean disc area is derived from the average of three orthogonal transthoracic echocardiography measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Liuliu Huang, MD, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) would not be shared, according to local authority data privacy policy.